CLINICAL TRIAL: NCT02011243
Title: Evaluation of the Internal Rotation Deficit of the Glenohumeral Joint in Advanced-level Handball Players Occurring Over One Training Season
Brief Title: Internal Rotation Deficit of the Glenohumeral Joint in Advanced-level Handball Players
Acronym: GIRDH
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2013/OM-01; 2013-A01183-42 (Other: RCB number)
Record Dates: First submitted 2013-12-09; First posted 2013-12-13 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Internal Rotation Contracture-shoulder; Articulation Disorders; Athletic Injuries
Keywords: deficit; internal rotation; gleno humeral articulation; hand ball
MeSH Terms: conditions — Articulation Disorders; Athletic Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Professional players, men: This group includes professional, male, handball players meeting study inclusion criteria.
- Professional players, women: This group includes professional, female, handball players meeting study inclusion criteria.
- Junior players, men: This group includes junior, male, handball players meeting study inclusion criteria.
- Junior players, women: This group includes junior, female, handball players meeting study inclusion criteria.

SUMMARY:
The main objective of this study is to estimate the incidence and prevalence of Internal Rotation Deficit (IRD) defined by a measure of IRD 2 (Internal Rotation Deficit in position 2) strictly greater than 20 ° in a population of advanced-level handball players over a training season.

DETAILED DESCRIPTION:
The secondary objectives of this study are :

A- To estimate and compare the prevalence of Internal Rotation Deficit within groups

B- To assess the association between the Internal Rotation Deficit and the appearance of a shoulder pain and/or discomfort when throwing

C- To assess the association between Internal Rotation Deficit and the appearance of a shoulder pathology demonstrated by clinical examination by at least one abnormality in one of the following three tests: the arming apprehension test, the relocation test or the O'Brien test

D- Assess changes in values of IRD 2, the ratio IRD 2/GRE 2, and the Total Range of Motion over the training season

E- Evaluate the association between the values of IRD 2 and the appearance of shoulder pain or discomfort when throwing

F- To evaluate the association between IRD 2 values and the appearance of a shoulder pathology (at least one anomaly in one of three tests: the arming apprehension test, the relocation test or the O'Brien test).

G- To assess the association between values of the IRD 2/GRE 2 ratio and the appearance of shoulder pain or discomfort when throwing

H- To assess the association between values of the IRD 2/GRE 2 ratio and the appearance of a shoulder pathology (at least one anomaly in one of three tests: the arming apprehension test, the relocation test or the O'Brien test).

I- To estimate the optimal threshold value of the IRD 2/GRE 2 ratio that would define an Internal Rotation Deficit in a more relevant fashion as compred to the IRD 2 alone

ELIGIBILITY:
Inclusion Criteria:

* The subject or his/her legal guardian must have given his/her informed and signed consent
* The subject must be insured or beneficiary of a health insurance plan
* The subject is a member of the professional and pre-professional handball clubs in Nîmes, France (the USAM or HBCN clubs) -- OR-- a member of the training centers associated with the same clubs whose parents or legal representatives have given informed consent

Exclusion Criteria:

* The subject is under judicial protection, under tutorship or curatorship
* The subject or his/her legal respresentative refuses to sign the consent
* It is impossible to correctly inform the subject
* The subject is pregnant, parturient, or breastfeeding
* The subject has been operated for shoulder instability, regardless of the surgical technique used
* The subject has a history of fracture of the proximal end of the humerus and / or elbow
* The subject has a history of rotator cuff surgery
* The subject has neurological or spinal problems, or has received physiotherapy on the shoulder complex within 30 days prior to the study assessment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population is composed of all members of the professional and pre-professional handball clubs in the city of Nîmes, France (the USAM and HBCN clubs). Younger players who are members of the training centers associated with these same clubs will also be included.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2014-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Presence/absence of an internal rotation deficit (IRD 2 > 20°) | 6 months
  IRD 2 = internal rotation deficit in position 2 Position 2 = dominant arm in abduction at 90°

SECONDARY OUTCOMES:
Presence/absence of an internal rotation deficit (IRD 2 > 20°) | baseline (Day 0)
Presence/absence of an internal rotation deficit (IRD 2 > 20°) | 3 months
Measure of the internal rotation deficit | baseline (day 0)
Measure of the internal rotation deficit | 3 months
Measure of the internal rotation deficit | 6 months
The ratio of DRI 2 / GRE 2 | baseline (day 0)
  GRE 2 = measure of the external gain in rotation in position 2 Position 2 = dominant arm in abduction at 90°
The ratio of DRI 2 / GRE 2 | 3 months
The ratio of DRI 2 / GRE 2 | 6 months
Measure of the total range of motion | baseline (day 0)
Measure of the total range of motion | 3 months
Measure of the total range of motion | 6 months
Presence/absence of pain when throwing (yes/no) | baseline (day 0)
Presence/absence of pain when throwing (yes/no) | 3 months
Presence/absence of pain when throwing (yes/no) | 6 months
Presence of discomfort when throwing (visual analog scale from 0 to 100) | baseline (day 0)
Presence of discomfort when throwing (visual analog scale from 0 to 100) | 3 months
Presence of discomfort when throwing (visual analog scale from 0 to 100) | 6 months
Presence/absence of shoulder pathology | baseline (day 0)
Presence/absence of shoulder pathology | 3 months
Presence/absence of shoulder pathology | 6 months
Shoulder clinical exam: the arming apprehension test | baseline (day 0)
Shoulder clinical exam: the arming apprehension test | 3 months
Shoulder clinical exam: the arming apprehension test | 6 months
Shoulder clinical exam: relocation test | baseline (day 0)
Shoulder clinical exam: relocation test | 3 months
Shoulder clinical exam: relocation test | 6 months
Shoulder clinical exam: the O'Brien test | baseline (day 0)
Shoulder clinical exam: the O'Brien test | 3 months
Shoulder clinical exam: the O'Brien test | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Marès, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France